CLINICAL TRIAL: NCT01471132
Title: Phase 2 Study of Sequential Hyperthermic Intraperitoneal Chemotherapy of Oxaliplatin and Paclitaxel for Gastric Cancer Patients With Peritoneum Metastasis or Positive Free Cancer Cells in Abdomen
Brief Title: Sequential HIPEC of Oxaliplatin and Paclitaxel for Gastric Cancer Patients With Peritoneum Metastasis
Acronym: SHOP-G01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-GCOT
Record Dates: First submitted 2011-11-01; First posted 2011-11-11 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Gastric Cancer; Metastases to Perineum
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 345mg/m2,43℃，30mins
Drug: Paclitaxel — Paclitaxel 260mg/m2,43℃，30mins

SUMMARY:
The recurrence and metastasis of peritoneum is always the lethal consequence for gastric cancer patients, and there is no effective therapy until now. It has been reported by Dr.Fujimoto that intraperitoneal chemotherapy plus hyperthermic therapy, which called hyperthermic intraperitoneal chemotherapy (HIPEC), can eliminate and suppress the free cancer cells and tiny metastasis in abdomen. Refer to the experience of systematic chemotherapy, HIPEC with combination regimen would have a brighter prospect. In this study, the investigators would use Oxaliplatin and paclitaxel sequent as HIPEC regimen. The safety and overall survival would be observed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved gastric adenocarcinoma.
* Peritoneum metastasis is observed or suspected by laparoscopy or radiologic examination,or free cancer cells are detected in peritoneal lavage liquid.
* Potentially resectable gastric cancer.
* ALT, AST < 80U/L; Total Bilirubin < 30μmol/L; WBC > 4x10^9/L; PLT > 100x10^9/L; Cr < 1.5 fold normal value.
* ECOG 0-2 points.
* Expected survival time longer than 3 months.
* Informed consent.

Exclusion Criteria:

* Recurrent gastric cancer.
* Pregnant or lactating women.
* Allergic to oxaliplatin or paclitaxel.
* Abnormal liver/kidney function.
* Serious heart/metabolic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | every 3 month postoperation up to 24 months

SECONDARY OUTCOMES:
Safety | every 3 month postoperation up to 24 months
  Number of Participants with Adverse Events(III or IV grades according to NCI-CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China